CLINICAL TRIAL: NCT07129785
Title: Dynamic Surface Exercise Training and Static Surface Exercise Training in Cerebral Palsy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Iqra Rashid, Student, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB/25/09/0036
Record Dates: First submitted 2025-08-11; First posted 2025-08-19 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Cerebral Palsy (CP); Spastic Diplegia Cerebral Palsy; Gross Motor Functions; Balance
Keywords: Dynamic Surface Exercise Training; Static Surface Exercise Training; Swiss Ball Therapy; Pediatric Neurorehabilitation; Postural Control; Gross Motor Function Measure; Pediatric Balance Scale; Trunk Control; Motor Skill Development; Unstable Surface Training; Stable Surface Training
MeSH Terms: conditions — Cerebral Palsy; Cerebral palsy, spastic, diplegic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic Surface Exercise Training (DSET) (Experimental): Participants in this group will receive Dynamic Surface Exercise Training for 60 minutes per session, four days per week, for six weeks. Activities include optimal arousal (active/passive bouncing) on Swiss/gym balls or trampolines, multi-planar trunk activation, high sitting with one- and two-hand reaching, sit-to-stand transitions, and dynamic balance tasks performed on unstable surfaces such as bolsters and platform swings. Exercises are designed to challenge vestibular, proprioceptive, and visual systems to enhance gross motor function and balance.
  Interventions: Behavioral: Dynamic Surface Exercise Training (DSET)
- Static Surface Exercise Training (SSET) (Active Comparator): Participants in this group will receive Static Surface Exercise Training for 60 minutes per session, four days per week, for six weeks. Activities include transfers between sitting and quadruped, high sitting on a bench with functional reaching, static and dynamic balance in standing, ball-catching and kicking, and trunk activation tasks performed on stable surfaces such as mats or benches. Exercises aim to improve gross motor function and balance through controlled, stable postural activities.
  Interventions: Behavioral: Static Surface Exercise Training (SSET)

INTERVENTIONS:
Behavioral: Dynamic Surface Exercise Training (DSET) — DSET involves performing multi-planar trunk activation, postural control, and balance exercises on unstable surfaces such as Swiss/gym balls, bolsters, trampolines, and platform swings. Each session lasts 60 minutes, four times per week, for six weeks. Activities include optimal arousal (bouncing), high sitting with one- and two-hand reaching, sit-to-stand transitions, and lateral weight-shifting. The unstable surface provides postural perturbations that stimulate vestibular, proprioceptive, and visual systems to improve gross motor function and balance in children with spastic diplegic cerebral palsy.
  Arms: Dynamic Surface Exercise Training (DSET)
Behavioral: Static Surface Exercise Training (SSET) — SSET consists of functional strength, posture, and balance exercises performed on stable surfaces such as mats, benches, or stools. Each session lasts 60 minutes, four times per week, for six weeks. Activities include transfers between sitting and quadruped, high sitting with functional reaching, static and dynamic standing balance, ball-catching and kicking, and trunk activation tasks. Exercises aim to enhance gross motor function and balance through controlled, stable postural activities in children with spastic diplegic cerebral palsy.
  Arms: Static Surface Exercise Training (SSET)

SUMMARY:
This randomized clinical trial aims to compare the effects of Dynamic Surface Exercise Training (DSET) and Static Surface Exercise Training (SSET) on balance and gross motor function in children with spastic diplegic cerebral palsy (CP) aged 6-12 years, classified at Gross Motor Function Classification System (GMFCS) levels III-IV. CP is the most common motor disability of childhood, characterized by non-progressive disturbances to the developing brain, leading to impairments in movement, posture, and functional independence. Balance deficits and gross motor limitations significantly impact daily activities and quality of life in these children.

Dynamic surfaces such as Swiss balls, bolsters, and platform swings provide postural perturbations that challenge vestibular, proprioceptive, and visual systems, potentially enhancing trunk control, postural stability, and adaptive responses. In contrast, static surface exercises emphasize controlled strength, postural alignment, and functional task performance on stable platforms such as mats or benches.

Fifty participants meeting the inclusion criteria will be randomly allocated into two equal groups. The DSET group will receive 60-minute sessions, four days per week for six weeks, involving multi-planar trunk activation, optimal arousal activities, and dynamic balance tasks on unstable surfaces. The SSET group will perform equivalent-duration exercises on stable surfaces, focusing on functional reaching, transfers, and static/dynamic balance.

Primary outcomes are Gross Motor Function Measure-66 (GMFM-66) and Pediatric Balance Scale (PBS), assessed at baseline, week 3, and week 6 by a blinded evaluator. Statistical analyses will compare within- and between-group changes. Findings will help identify the more effective approach for improving functional outcomes in children with CP, guiding evidence-based pediatric neurorehabilitation strategies.

DETAILED DESCRIPTION:
Cerebral palsy (CP) encompasses a group of permanent disorders affecting movement and posture due to non-progressive disturbances in the developing fetal or infant brain. Spastic diplegic CP often results in muscle tone abnormalities, postural instability, and reduced gross motor function. These impairments hinder participation in daily activities and increase fall risk. Motor deficits are closely linked to postural control, which depends on integrated sensory input from visual, vestibular, and somatosensory systems.

Dynamic surface training introduces controlled instability through tools like Swiss balls, bolsters, trampolines, and platform swings. This variability promotes adaptive postural adjustments and multi-planar muscle activation, potentially enhancing gross motor skills and balance beyond what is achieved with stable surfaces. Static surface training, using mats, benches, or floors, emphasizes strength, posture, and functional movement without additional instability challenges.

This single-center, single-blinded, randomized clinical trial will recruit 50 children aged 6-12 years with spastic diplegic CP (GMFCS III-IV) who can follow verbal commands and meet other inclusion criteria. Participants will be randomly allocated to:

Group A (DSET): 6-week program, 60 min/day, 4 days/week. Activities include optimal arousal (active/passive bouncing), high sitting with one-hand/both-hands reaching, sit-to-stand transitions, multi-directional reaching, trunk activation, and dynamic balance exercises on unstable surfaces.

Group B (SSET): 6-week program, 60 min/day, 4 days/week. Exercises include transfers between sitting and quadruped, high sitting on a bench with functional reaching, static/dynamic standing balance, and trunk activation tasks on stable surfaces.

Outcome Measures:

Primary: GMFM-66 (gross motor function), PBS (balance performance).

Secondary: Functional improvement trends over time.

Assessments will occur at baseline, week 3, and week 6, conducted by blinded assessors. Data will be analyzed using SPSS v24, applying parametric or non-parametric tests based on data normality, with significance set at p ≤ 0.05.

Ethical approval has been obtained from the Institutional Research Ethics Board of the University of Lahore. Written informed consent will be obtained from parents/guardians. Participant confidentiality will be maintained, and participation will be voluntary.

The study is designed to address gaps in existing literature, including limited sample sizes, lack of long-term follow-up, and variability in intervention protocols. Results will provide clinically relevant evidence on whether unstable or stable surface training is more effective for improving motor function and balance in children with spastic diplegic CP, supporting optimized rehabilitation planning.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with spastic diplegic CP between age 6-12 years (Reddy & Balaji, 2020).
* Both male and female gender (Reddy & Balaji, 2020).
* Who were able to follow verbal commands.
* Children having level III and IV of Gross Motor Function Classification System (GMFCS) (Reddy & Balaji, 2020).

Exclusion Criteria:

* CP Child who were reluctant to cooperate.
* CP child having visual or intellectual impairments (Reddy & Balaji, 2020).
* Who were on Antiepileptic medications (Reddy & Balaji, 2020).
* CP child having any cardiac or chest anomalies and hearing deficits.
* Exercise intolerance and any recent orthopedic surgery will also be excluded from the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure-66 (GMFM-66) Score | Baseline, Week 3, Week 6
  The GMFM-66 is a standardized observational instrument used to assess gross motor function in children with cerebral palsy. It evaluates the child's ability to perform various motor tasks across lying, sitting, crawling, standing, and walking dimensions. Scores range from 0 to 100, with higher scores indicating better motor performance. Assessments will be conducted by a blinded evaluator at baseline, week 3, and week 6 to determine within- and between-group changes following Dynamic Surface Exercise Training or Static Surface Exercise Training.
Pediatric Balance Scale (PBS) Score | Baseline, Week 3, Week 6
  The PBS is a 14-item scale adapted from the Berg Balance Scale to assess static, dynamic, and functional balance in children aged 3-13 years. Each item is scored from 0 to 4, with total scores ranging from 0 to 56. Higher scores reflect better balance and postural control. A blinded evaluator will assess participants at baseline, week 3, and week 6 to measure improvement in balance performance after the assigned intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No